CLINICAL TRIAL: NCT02470299
Title: A Randomized Placebo-controlled Evaluation of GTPase Inhibition by Post-operative Intravenous Ketorolac in Ovarian Cancer Patients
Brief Title: Evaluation of GTPase Inhibition by Post-operative Intravenous Ketorolac in Ovarian Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: INST 1420
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: ketorolac; GTPase; cancer; peritoneal; fallopian; ovarian
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Neoplasms | interventions — Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketorolac (Experimental): Once deemed stable in the first 1-3 post-operative days, patients will be receive age-based ketorolac (30 mg <65, 15mg > 65) daily for three days
  Interventions: Drug: Ketorolac
- Placebo (Placebo Comparator): Once deemed stable in the first 1-3 post-operative days, patients will be receive placebo daily for three days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ketorolac — Ketorolac tromethine 15 mg or 30 mg doses will be administered via intravenous (IV) push undiluted over 15 - 30 seconds
  Ketorolac will be dosed according to FDA approved recommendations. For planned three daily dose (IV) based on clinical scenario:
  * Patients < 65 years of age: Daily dose of 30 mg for three doses.
  * Patients ≥ 65 years of age, renally impaired and/or less than 50 kg (110 lbs) of body weight: Daily dose of 15 mg for three doses
  Blood and peritoneal fluid will be drawn prior to each dose (time 0, 24, 48, 72 hr) as well as at 6 hr after the first dose
  Other Names: Toradol
  Arms: Ketorolac
Other: Placebo — Equivalent volume of normal saline will be set in the syringe for each daily dose registered for the patient in a blinded fashion. The volume will be determined by the dose calculation as follows: For planned three daily dose (IV) based on clinical scenario:
  * Patients < 65 years of age: Daily dose of 30 mg for three doses.
  * Patients ≥ 65 years of age, renally impaired and/or less than 50 kg (110 lbs) of body weight: Daily dose of 15 mg for three doses.
  Blood and peritoneal fluid will be drawn prior to each dose (time 0, 24, 48, 72 hr) as well as at 6 hr after the first dose
  Arms: Placebo

SUMMARY:
There is a move towards personalized medicine in cancer care, and significant effort is underway to evaluate new targeted therapeutics for the treatment of ovarian cancer. One way to identify potential new drug targets is by screening a drug library to determine whether drugs in the library target key kinase or enzymatic sites in cellular signaling pathways. Previous preclinical work and pilot studies demonstrated that ketorolac (a type of non-steroidal anti-inflammatory drug) inhibits GTPase activity in ovarian cancer cells retrieved from the post-operative peritoneal cavity.

The purpose of this study is to confirm that this inhibitory effect is ketorolac driven and not a specific effect of the post-operative peritoneal compartment.

DETAILED DESCRIPTION:
Drug repurposing, screening a library of FDA approved agents, can identify agents that are clinically available and for which pharmacology and pharmacokinetics are known and preclinical data can be generated rapidly without the subsequent need for GMP (good manufacturing practice) new drug production. Small GTPases, including members of the Rab, Ras and Rho families, are attractive targets for the development of cancer therapeutics based on their pivotal roles in protein trafficking, proliferation/survival and cytoskeletal organization, respectively. Ketorolac tromethamine is a non-steroidal anti-inflammatory drug that was identified in previous in-silico drug screens to be an inhibitor of GTPases. In a previous phase 0 clinical study, ketorolac was administered intravenously to ovarian cancer patients following optimal cytoreductive surgery. Ovarian cancer cells were obtained at the time of surgery, prior to ketorolac administration, and at various times after ketorolac dosing. Analysis of GTPase activity in these specimens showed a time-dependent inhibition of Rac1 and Cdc42 GTPase activity. The purpose of this study is to confirm that the effect is ketorolac driven and not a specific effect of the post-operative peritoneal compartment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be suspected of having a diagnosis of ovarian, fallopian tube or primary peritoneal cancer with a planned cytoreductive surgery.
* Borderline ovarian cancer with ascites is allowable.
* ECOG/Zubrod/SWOG Performance Status <2 (Karnofsky Performance Status > 70%)
* Female' age ≥18 years
* Ability to provide informed consent
* Baseline laboratory values (bone marrow, renal, hepatic):

  * Adequate bone marrow function:

    * Absolute neutrophil count >1000/µL
    * Platelet count >100'000/µL
  * Renal function:

    * Serum creatinine < 1.5 x ULN
  * Hepatic function:

    * Bilirubin <1.5x normal
    * Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamic-pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) levels ≤ 2 x ULN
* No known bleeding disorders
* No known sensitivity or allergy to NSAIDs
* No active peptic ulcer disease
* No active bleeding

Secondary Eligibility

* Histologic diagnosis of epithelial ovarian, fallopian tube or primary peritoneal cancer confirmed on frozen section diagnosis during debulking surgery
* Attempted maximal cytoreductive surgery. Patients will still be eligible whether optimal or suboptimally debulked at the completion of the surgery.
* No active bleeding in the post-operative period

Exclusion Criteria:

* Non-epithelial ovarian cancer or metastatic cancer from another site to the ovaries
* Borderline ovarian cancer without ascites
* Uncontrolled or unstable medical conditions
* Off study use of ketorolac or other NSAIDs prior to study administration within the perioperative window (7 days before surgery and up to the time of planned study administration)
* Active bleeding or high risk of bleeding
* Active therapeutic anticoagulation
* Known hypersensitivity to NSAIDs
* Chronic or acute renal insufficiency as defined by a preoperative serum creatinine greater than 1.5 mg/dL or creatinine clearance of < 40 ml/min
* Any co-morbid condition that' in the view of the attending physician' renders the patient at high risk from ketorolac treatment complications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-10-29 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Ketorolac inhibition of GTPase activity | Within 4 weeks of peritoneal cell collection
  Ovarian cancer cells retrieved from the post-debulked peritoneal cavity after three intravenous dosings of ketorolac will be evaluated for GTPase activity using cell-based laboratory assays

SECONDARY OUTCOMES:
Intraperitoneal and serum pharmacokinetics of ketorolac | Within 4 weeks of peritoneal and blood specimen collection
  Serum and intraperitoneal concentrations of ketorolac will be assessed over time using high performance liquid chromatography (HPLC)
Time to CA-125 normalization | Up to 6 months following first ketorolac treatment
  CA-125 will be measured using a standard laboratory assay
Toxicity assessment | Up to 30 days following first ketorolac treatment
  Subjective/objective evidence of developing drug toxicity will be evaluated according to NCI-CTC toxicity criteria (CTCAE version 3.0)

OTHER OUTCOMES:
Overall survival (Exploratory objective) | Up to 5 years following first ketorolac treatment
  Time from treatment to death due to any cause
Progression free survival (Exploratory objective) | Up to 18 months following first ketorolac treatment
  Time from treatment to progressive disease or death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Y. Muller, MD, Principal Investigator — University of New Mexico Comprehensive Cancer Center
Locations (1):
- Universtiy of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No